CLINICAL TRIAL: NCT01198197
Title: PET Brain and Whole Body Distribution Studies for Nociceptin/Orphanin FQ Peptide (NOP) Receptor Using [(11)C]NOP-1A
Brief Title: PET Brain and Whole Body Distribution Studies for Nociceptin/Orphanin FQ Peptide (NOP) Receptor Using [11C]NOP-1A
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100204; 10-M-0204
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-09-05

CONDITIONS: Pain; Anxiety; Depression
Keywords: Nociceptin/Orphanin FQ Peptide (NOP); PET Imaging; Brain Imaging; Healthy Volunteer; HV
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression | interventions — 3-(2'-fluoro-6',7'-dihydrospiro(piperidine-4,4'-thieno(3,2-c)pyran)-1-yl)-2-(2-fluorobenzyl)-N-methylpropanamide

INTERVENTIONS:
Drug: NOP-1A

SUMMARY:
Background:

- A small brain protein called nociceptin/orphanin FQ peptide (NOP) receptor may be involved in several brain diseases such as anxiety, depression, drug abuse, and seizures. Researchers are interested in testing a new radioactive chemical that will help locate NOP receptors in the brain during imaging studies such as positron emission tomography (PET) scans. Because this chemical has not yet been approved by the Food and Drug Administration, it is considered to be an experimental drug.

Objectives:

- To investigate the effectiveness of the experimental chemical [11C]NOP-1A in imaging studies of the nociceptin/orphanin FQ peptide (NOP) receptor.

Eligibility:

- Healthy volunteers between 18 and 50 years of age who are able to have imaging studies.

Design:

* This study will involve three or four outpatient visits to the National Institutes of Health Clinical Center. All participants will be screened with a full physical examination, medical history, blood and urine tests, and electrocardiogram.
* Participants will be involved in one or more parts of this three-part study as directed by study researchers. Part 1 consists of brain imaging to study how the brain responds to the chemical. Part 2 is a whole body imaging study to evaluate how the chemical is distributed throughout the body after being administered. Part 3 is a set of testing and retesting scans to determine how precise the drug is in locating the NOP receptors in the brain.
* Part 1: Participants will have a brain magnetic resonance imaging (MRI) scan. Then the study drug will be administered and participants will have a brain PET scan. Blood samples will be taken during the PET scan, and urine samples will be taken after the scan. These tests will take up to 3 hours to perform.
* Part 2: Participants will have a whole body PET scan that will last a maximum of 3 hours.
* Part 3: Participants will receive the study drug and have two additional PET scans. Blood samples will also be taken during this part.

DETAILED DESCRIPTION:
Nociceptin/orphanin FQ peptide (NOP) receptor is a new class of opioid receptor cloned in 1994 before identifying the endogenous ligand. Within a year, endogenous ligand was identified and soon many ligands were developed and evaluated in vitro and in vivo for NOP receptor distribution and activity. NOP receptor is widely distributed in brain, spinal cord and in peripheral organs such as heart, lungs, kidney, intestine and liver. Being a G-protein coupled receptor, its activation leads to changes in intracellular signal transduction mediated by adenylyl cyclase, Ca(2+) and K(+) ion channels, mitogen-activated kinase and phospholipase C. Based on preclinical studies, NOP receptor is implicated in regulation of pain, anxiety and depression, drug abuse, feeding, learning/memory, and motor activity.

Since the time of cloning the receptor and identification of endogenous ligand, numerous compounds have been designed targeting this receptor. However, there are no PET radioligands currently available to study NOP distribution and activity in humans. We wish to test a newly developed PET radioligand, [(11)C]NOP-1A to study the role of NOP receptors in humans.

The purpose of this protocol is (1) to perform brain imaging using [(11)C]NOP-1A in healthy volunteers to characterize the brain uptake and distribution (2) to perform whole body PET studies in healthy volunteers in order to estimate radiation absorbed doses for [(11)C]NOP-1A, (3) to perform brain test-retest studies in healthy volunteers in order to further examine the precision of the measurement of receptor binding and to determine optimal parameters for future experiments using [(11)C]NOP-1A, and, (4) to compare [(11)C]NOP-1A concentrations in artery and vein of healthy volunteers to assess the feasibility of replacing the arterial line with a less invasive venous line for brain scans.

Successful development of a PET radioligand to image NOP receptor will have a strong impact on further understanding and clinical management of neuropsychiatric disorders that are mediated by opioid receptor system. Future experiments will include studies on any relevant neuropsychiatric disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers:

Subjects must be adults between 18-50 years old.

Subjects must be able and willing to give written informed consent.

EXCLUSION CRITERIA:

Current psychiatric illness or severe systemic disease based on history and physical exam.

If women, pregnancy or breast feeding (betaHCG will be measured in all female patients within 24 hours of scan and must be negative)

Clinically significant laboratory abnormalities.

Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases or any cardiopulmonary disease.

Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.

Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.

Positive urine drug screen at screening.

Inability to lie flat on camera bed for about 2.5 hours

Subjects who have metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-09-03; Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
For the PET scans, we will measure the regional densities of NOP receptors as distribution volume (VT). Distribution volume is the ratio at equilibrium of brain uptake to the concentration of parent radioligand in plasma. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berthele A, Platzer S, Dworzak D, Schadrack J, Mahal B, Buttner A, Assmus HP, Wurster K, Zieglgansberger W, Conrad B, Tolle TR. [3H]-nociceptin ligand-binding and nociceptin opioid receptor mrna expression in the human brain. Neuroscience. 2003;121(3):629-40. doi: 10.1016/s0306-4522(03)00484-6. PMID 14568023
- [Background] Bridge KE, Wainwright A, Reilly K, Oliver KR. Autoradiographic localization of (125)i[Tyr(14)] nociceptin/orphanin FQ binding sites in macaque primate CNS. Neuroscience. 2003;118(2):513-23. doi: 10.1016/s0306-4522(02)00927-2. PMID 12699786
- [Background] Brown AK, Fujita M, Fujimura Y, Liow JS, Stabin M, Ryu YH, Imaizumi M, Hong J, Pike VW, Innis RB. Radiation dosimetry and biodistribution in monkey and man of 11C-PBR28: a PET radioligand to image inflammation. J Nucl Med. 2007 Dec;48(12):2072-9. doi: 10.2967/jnumed.107.044842. Epub 2007 Nov 15. PMID 18006619